CLINICAL TRIAL: NCT03530436
Title: Comparison of the Bioavailability of Different Curcumin Formulations in Healthy Humans
Brief Title: Comparison of Curcumin Bioavailability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HS-CUV-2018
Record Dates: First submitted 2018-04-25; First posted 2018-05-21 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Safety After Oral Intake; Pharmacokinetics After Oral Intake
Keywords: Bioavailability; Pharmacokinetics; Curcumin; Demethoxycurcumin; Bisdemethoxycurcumin
MeSH Terms: interventions — turmeric extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Native turmeric extract (Other): 6 capsules of native curcumin (207 mg curcumin)
  Interventions: Dietary Supplement: Native turmeric extract
- Native turmeric extract with 7-9% volatile turmeric oils (Experimental): 6 capsules of the formulation; dosage normalized to 207 mg curcumin
  Interventions: Dietary Supplement: Native turmeric extract with 7-9% volatile turmeric oils
- Turmeric extract plus mixture of phytochemicals (Experimental): 6 capsules of the formulation; dosage normalized to 207 mg curcumin
  Interventions: Dietary Supplement: Turmeric extract plus mixture of phytochemicals
- Cyclodextrin complex of curcuminoids (Experimental): 6 capsules of the formulation; dosage normalized to 207 mg curcumin
  Interventions: Dietary Supplement: Cyclodextrin complex of curcuminoids
- Turmeric oleoresin (Experimental): 6 capsules of the formulation; dosage normalized to 207 mg curcumin
  Interventions: Dietary Supplement: Turmeric oleoresin
- Liposomal curcumin (Experimental): 6 capsules of the formulation; dosage normalized to 207 mg curcumin
  Interventions: Dietary Supplement: Liposomal curcumin
- Phytosomal curcumin (Experimental): 6 capsules of the formulation; dosage normalized to 207 mg curcumin
  Interventions: Dietary Supplement: Phytosomal curcumin
- Micellar turmeric extract (Experimental): 6 capsules of the formulation; dosage normalized to 207 mg curcumin
  Interventions: Dietary Supplement: Micellar turmeric extract

INTERVENTIONS:
Dietary Supplement: Native turmeric extract — 207 mg curcumin
  Arms: Native turmeric extract
Dietary Supplement: Native turmeric extract with 7-9% volatile turmeric oils — 207 mg curcumin
  Arms: Native turmeric extract with 7-9% volatile turmeric oils
Dietary Supplement: Turmeric extract plus mixture of phytochemicals — 207 mg curcumin
  Arms: Turmeric extract plus mixture of phytochemicals
Dietary Supplement: Cyclodextrin complex of curcuminoids — 207 mg curcumin
  Arms: Cyclodextrin complex of curcuminoids
Dietary Supplement: Turmeric oleoresin — 207 mg curcumin
  Arms: Turmeric oleoresin
Dietary Supplement: Liposomal curcumin — 207 mg curcumin
  Arms: Liposomal curcumin
Dietary Supplement: Phytosomal curcumin — 207 mg curcumin
  Arms: Phytosomal curcumin
Dietary Supplement: Micellar turmeric extract — 207 mg curcumin
  Arms: Micellar turmeric extract

SUMMARY:
The curcuminoids curcumin, demethoxycurcumin and bisdemethoxycurcumin can be found in the rhizome of turmeric (Curcuma longa). Curcumin is widespread used for colouring foods. Based on its natural low bioavailability and the number of its effects on human health, several approaches such as increasing its water solubility or inhibiting its metabolism were taken to improve its bioavailability. Pharmacokinetics of curcumin from various supplements using those different mechanisms have been compared to the one of native curcumin. The investigator's study here will compare the bioavailability of curcumin from eight different curcumin formulations with native curcumin and between themselves. The study will folllow a single dose (in form of curcumin formulations, normalized to 207 mg curcumin), placebo-controlled, randomized, double-blind, nine-armed crossover study design with ≥ 1-week washout periods. Plasma samples will be collected at intervals up to 24 hours after intake. Investigators will compare the pharmacokinetics between the different curcumin formulations and to native curcumin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers with blood chemistry values within normal ranges
* Body mass index in a normal range

Exclusion Criteria:

* Pregnancy or lactation
* Alcohol and or drug abuse
* Use of dietary supplements or any medications except contraceptives
* Any known malignant, metabolic and endocrine diseases
* Previous cardiac infarction
* Dementia
* Blood pressure >140/90 mmHg
* Resting heart rate not within 50 to 90 beats per minute
* Participation in a clinical trial within the past 6 weeks
* Smoking
* Physical activity of more than 5 h per wk

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Mean area under the curve (AUC) of plasma concentration vs. time of total curcumin [nmol/L*h] | 0, 1, 2, 4, 6, 8 and 24 hours post dose
  Total curcumin after deconjugation with β-glucuronidase
Mean area under the curve (AUC) of plasma concentration vs. time of total demethoxycurcumin [nmol/L*h] | 0, 1, 2, 4, 6, 8 and 24 hours post dose
  Total demethoxycurcumin after deconjugation with β-glucuronidase
Mean area under the curve (AUC) of plasma concentration vs. time of total bisdemethoxycurcumin [nmol/L*h] | 0, 1, 2, 4, 6, 8 and 24 hours post dose
  Total bisdemethoxycurcumin after deconjugation with β-glucuronidase
Maximum plasma concentration (Cmax) of total curcumin [nmol/L] | 0, 1, 2, 4, 6, 8 and 24 hours post dose
  Total curcumin after deconjugation with β-glucuronidase
Maximum plasma concentration (Cmax) of total demethoxycurcumin [nmol/L] | 0, 1, 2, 4, 6, 8 and 24 hours post dose
  Total demethoxycurcumin after deconjugation with β-glucuronidase
Maximum plasma concentration (Cmax) of total bisdemethoxycurcumin [nmol/L] | 0, 1, 2, 4, 6, 8 and 24 hours post dose
  Total bisdemethoxycurcumin after deconjugation with β-glucuronidase
Time to reach maximum plasma concentration (Tmax) of total curcumin [h] | 0, 1, 2, 4, 6, 8 and 24 hours post dose
  Total curcumin after deconjugation with β-glucuronidase
Time to reach maximum plasma concentration (Tmax) of total demethoxycurcumin [h] | 0, 1, 2, 4, 6, 8 and 24 hours post dose
  Total demethoxycurcumin after deconjugation with β-glucuronidase
Time to reach maximum plasma concentration (Tmax) of total bisdemethoxycurcumin [h] | 0, 1, 2, 4, 6, 8 and 24 hours post dose
  Total bisdemethoxycurcumin after deconjugation with β-glucuronidase

CONTACTS AND LOCATIONS:
Overall Officials: Jan Frank, Prof. Dr., Principal Investigator — University of Hohenheim
Locations (1):
- University of Hohenheim, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the research group — http://www.nutrition-research.de/